CLINICAL TRIAL: NCT03490318
Title: Effectiveness of Multimodal Imaging for the Evaluation of Retinal Oedema And New vesseLs in Diabetic Retinopathy
Acronym: EMERALD
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17020NL-AS; 10856638 (Registry Identifier: ISRCTN); 17/NI/0124 (Other: ORECNI)
Record Dates: First submitted 2017-12-05; First posted 2018-04-06 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Proliferative Diabetic Retinopathy; Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with DMO and/or PDR

SUMMARY:
Given the high number of people with DMO and PDR, the need for patients to be seen at short follow-up intervals, the need for frequent treatments and the requirement for long-term follow-up, there is a very large workload in Hospital Eye Services related to DMO/PDR which is making it difficult for the NHS to cope with the demand, in particular, due to shortage of ophthalmologists. This is only expected to get worse given the increasing prevalence of DM. Identifying new ways of increasing the NHS capacity and efficiency without compromising the quality of care would greatly benefit the NHS.

The purpose of this study is to determine whether successfully treated patients with DMO and PDR could be followed up without a face-to-face examination by an ophthalmologist. EMERALD will evaluate a new care pathway which will include multimodal retinal imaging and separate image assessment by trained ophthalmic graders. This new pathway will be compared to the current standard care pathway: for DMO: ophthalmologist evaluating patients in clinic by slit-lamp biomicroscopy and with access to OCT images; for PDR ophthalmologists evaluating patients in clinic by slit-lamp biomicroscopy. EMERALD will compare how accurate the new pathway is at determining which patients have active or inactive disease. The costs and acceptability of current and new models of care will also be compared.

DETAILED DESCRIPTION:
1. Research Hypothesis

   The hypothesis is that the new form of surveillance for people with stable DMO and/or PDR will be as sensitive as the current standard of care but at a lower cost.
2. Study Aim

   EMERALD aims to determine the diagnostic performance and cost-effectiveness of a new form of surveillance for people with stable DMO and/or PDR, using the current standard of care as the reference standard.
3. Study Objectives

The specific objectives of this study are to evaluate the new surveillance pathway to:

1. Quantify and compare the diagnostic accuracy (in terms of sensitivity, specificity, overall agreement, positive and negative likelihood ratios) of the new pathway of surveillance (ophthalmic grader pathway) using the current standard of care pathway as the reference standard. This will be done separately for DMO and PDR.
2. Assess acceptability of the new surveillance pathway.
3. Determine the proportion of patients requiring subsequent full clinical assessment by an ophthalmologist under the new pathway.
4. Determine the proportion of patients unable to undergo imaging tests, with images of inadequate quality and indeterminate findings under the new pathway.
5. Establish relative cost-effectiveness of the new surveillance pathway.

4. Outcome measures

4.1 Primary outcome

The primary outcome measure is:

• Sensitivity of the new pathway (ophthalmic grader pathway) in detecting active DMO/PDR, using the standard care pathway as the reference standard.

4.2 Secondary outcomes

There are a number of secondary outcomes which will be measured and include:

* Specificity, concordance (agreement) between new pathway (ophthalmic grader pathway) and the standard care pathway, positive and negative likelihood ratios
* Cost-effectiveness
* Acceptability
* Proportion of patients requiring subsequent full clinical assessment
* Proportions of patients unable to undergo imaging, with inadequate quality images or indeterminate findings.

  5. STUDY DESIGN

5.1 Study Design

EMERALD is a prospective, cross-sectional diagnostic study of patients with diabetic retinopathy and DMO or PDR (or both) who had been previously successfully treated and who, at the time of enrolment in the study, may have active or inactive disease (both are required to evaluate the diagnostic performance of the new pathway).

Specifically, EMERALD will have a case-referent cross-sectional diagnostic study design with both sampling (selection) of patients and data collection carried out prospectively (18). This approach provides both a cost-efficient study design while also having a low risk of bias in terms of diagnostic accuracy (19)

5.2 Study Setting

Specialist Hospital Eye Services (HES) in the UK. All centres involved have extensive experience with the management of patients with diabetic retinopathy, DMO and PDR.

6. End of Study

For the purposes of submitting the end of trial notification to the Sponsor and the Research Ethics Committee (REC), the end of trial will be considered to be when the database lock occurs for the final analysis. The trial will be stopped prematurely if:

* Mandated by the REC
* Mandated by the Sponsor (e.g. following recommendations from the Trial Steering Committee (TSC)
* Funding for the trial ceases The REC that originally gave a favourable opinion of the trial will be notified in writing when the trial has been concluded or if it is terminated early.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older) with type 1 or 2 diabetes with previously successfully treated DMO and/or PDR in one or both eyes and in whom, at the time of enrolment in the study, DMO and/or PDR may be active or inactive.
* Active DMO will be defined as a central subfield retinal thickness (CRT) of > 300 microns and/or presence of intraretinal/subretinal fluid on spectral domain OCT.
* Inactive DMO will be defined as no intraretinal/subretinal fluid
* Active PDR will be defined by the presence of sub-hyaloid/vitreous haemorrhage and/or active new vessels (new vessels with lack of fibrosis on them)
* Inactive PDR will be defined by the lack of preretinal/vitreous haemorrhage and lack of active new vessels.

Exclusion Criteria:

* Unable to provide informed consent
* Patients do not read, speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with type 1 or type 2 diabetes with previously successfully treated DMO and/or PDR and in whom, at the time of enrolment in the study, DMO and/or PDR may be active or inactive.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the new pathway (ophthalmic grader pathway) in detecting active DMO/PDR, using the standard care pathway as the reference standard. | 30 months
  Sensitivity analysis

SECONDARY OUTCOMES:
Specificity, concordance (agreement) between new pathway (ophthalmic grader pathway) and the standard care pathway, positive and negative likelihood ratios | 30 months
  specificity, concordance, positive and negative likelihood ratios
Cost-effectiveness | 30 months
  specificity analysis, QALY
Acceptability | 30 months
  specificity, concordance, positive and negative likelihood ratios
Proportion of patients requiring subsequent full clinical assessment | 30 months
  specificity, concordance, positive and negative likelihood ratios
Proportions of patients unable to undergo imaging, with inadequate quality images or indeterminate findings. | 30 months
  specificity, concordance, positive and negative likelihood ratios

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Lois, PhD, FRCS(Ed). FRCOphth., Principal Investigator — Queen's University, Belfast
Locations (13):
- United Kingdom (13):
  - James Cook University Hopsital, Middlesbrough, North Yorkshire
  - Queen Margaret Hospital, Dunfermline, Scotland
  - Royal Victoria Hospital, Belfast
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - Frimley Park Hospital, Frimley
  - Gloucestershire Royal Hospital, Gloucester
  - Moorfields eye Hospital, London
  - King's College Hospital, London
  - Manchester Eye Hospital, Manchester
  - Oxford John Radcliffe Hospital, Oxford
  - Sheffield Eye Hospital, Sheffield
  - City Hopsitals Sunderland, Sunderland

IPD SHARING:
Plan to Share IPD: Undecided
15.4 Data Sharing Statement
  Requests for data sharing will be reviewed on a case by case basis by the CI and TMG.
  15.5 Data Access
  Following the publication of the primary and secondary outcomes, there may be scope to conduct additional analyses on the data collected. In such instances, formal requests for data will need to be made in writing to the CI who will discuss this with the TMG. In the event of publications arising from such analyses, those responsible will need to provide the CI with a copy of any intended manuscript for approval prior to submission. Authorship will need to take the format of "[name] on behalf of the EMERALD Clinical Trial Group" or something similar, which will be agreed by the TMG.

REFERENCES:
- [Derived] Maredza M, Mistry H, Lois N, Aldington S, Waugh N; EMERALD Study Group. Surveillance of people with previously successfully treated diabetic macular oedema and proliferative diabetic retinopathy by trained ophthalmic graders: cost analysis from the EMERALD study. Br J Ophthalmol. 2022 Nov;106(11):1549-1554. doi: 10.1136/bjophthalmol-2021-318816. Epub 2021 Jun 3. PMID 34083209
- [Derived] Lois N, Cook J, Wang A, Aldington S, Mistry H, Maredza M, McAuley D, Aslam T, Bailey C, Chong V, Ghanchi F, Scanlon P, Sivaprasad S, Steel D, Styles C, Azuara-Blanco A, Prior L, Waugh N. Multimodal imaging interpreted by graders to detect re-activation of diabetic eye disease in previously treated patients: the EMERALD diagnostic accuracy study. Health Technol Assess. 2021 May;25(32):1-104. doi: 10.3310/hta25320. PMID 34060440
- [Derived] Lois N, Cook J, Aldington S, Waugh N, Mistry H, Sones W, McAuley D, Aslam T, Bailey C, Chong V, Ghanchi F, Scanlon P, Sivaprasad S, Steel D, Styles C, McNally C, Rice R, Prior L, Azuara-Blanco A; EMERALD Study Group. Effectiveness of Multimodal imaging for the Evaluation of Retinal oedema And new vesseLs in Diabetic retinopathy (EMERALD). BMJ Open. 2019 Jun 28;9(6):e027795. doi: 10.1136/bmjopen-2018-027795. PMID 31256030